CLINICAL TRIAL: NCT06676085
Title: A Novel Strategy Combined Regional Anticoagulation in Membrane Oxygenator and Low-intensity of Systemic Anticoagulation Applied in Management of Extracorporeal Membrane Oxygenation
Brief Title: A Novel Strategy of ECMO Management Using Nafamostat for Regional Combined With Low Intensity Systematic Anticoagulation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Nafamostat in ECMO
Record Dates: First submitted 2024-11-04; First posted 2024-11-06 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-10

CONDITIONS: ECMO
MeSH Terms: interventions — nafamostat; Heparin

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- New Anticoagulation Strategy Group (Experimental): Combination of nafamostat and unfractionated heparin for anticoagulation, adjusting the dosage of unfractionated heparin to maintain APTT in the body for 40-45 seconds, and adjusting the dosage of nafamostat to maintain APTT in the membranous lung for 50-60 seconds during ECMO
  Interventions: Drug: Nafamostat
- control group (Active Comparator): Anticoagulation with unfractionated heparin, regulating the dosage of unfractionated heparin to maintain APTT in the body for 50-60s during ECMO.
  Interventions: Drug: Heparin

INTERVENTIONS:
Drug: Nafamostat — Nafamostat combined with unfractionated heparin for anticoagulation
  Arms: New Anticoagulation Strategy Group
Drug: Heparin — unfractionated heparin for anticoagulation
  Arms: control group

SUMMARY:
ECMO is widely used in patients with refractory respiratory and/or circulatory failure.The data shows that the incidence of bleeding and thrombotic events is still above 40%,and it is closely related to the increase in mortality rate.Therefore, optimizing ECMO anticoagulation management to reduce bleeding and thrombotic events is a key scientific issue that urgently needs to be addressed.

ELIGIBILITY:
Inclusion Criteria:

* age older than 18 years old
* received ECMO because of severe respiratory failure

Exclusion Criteria:

* anticoagulant contraindications
* cerebral infarction or suspected patients
* severe hypertension
* women in gestational and lactational period
* hemophilia
* allergic to heparin or Nafamostat
* unwilling or unable to complete the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
incidence of ECMO related bleeding or thrombotic events | 28 days
  the incidence of ECMO related bleeding or thrombotic events,such as membrane oxygenator or tube thrombotic,local blooding.

CONTACTS AND LOCATIONS:
Overall Officials: Bing Sun, MD, Principal Investigator — Beijing Chao Yang Hospital
Locations (1):
- Bing Sun, Beijing, Beijing Municipality, China